CLINICAL TRIAL: NCT04623879
Title: Real Life Evaluation of the Multi-organ Effects of Lumacaftor/Ivacaftor on F508del Homozygous Cystic Fibrosis Patients.
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Karin Yaakobi Bianu, Senior physician, Pediatric Pulmonology Unit and CF Center, Carmel Medical Center
Other Study IDs: CMC-16-0108-CTIL
Record Dates: First submitted 2020-10-12; First posted 2020-11-10 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Cystic Fibrosis
Keywords: CFTR modulators; Lumacaftor/ Ivacaftor; Bone metabolism; Pancreatic function
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- F508del homozygous adult CF patients: F508del homozygous adult CF patients who commenced treatment with LUM-IVA
  Interventions: Drug: Lumacaftor, Ivacaftor Drug Combination

INTERVENTIONS:
Drug: Lumacaftor, Ivacaftor Drug Combination
  Other Names: Orkambi

SUMMARY:
Background: Lumacaftor/Ivacaftor (LUM-IVA), a CFTR corrector-potentiator combination, was found to improve lung function and reduce pulmonary exacerbations (PEx). However, cystic fibrosis (CF) is a multi-organ disease and therefore there is a need for more information on the systemic effects of CFTR modulators.

Aim: To evaluate pancreatic function, bone metabolism and respiratory changes through a year of LUM-IVA treatment.

Methods: A prospective real world, one-year study on F508del homozygous adult CF patients who commenced treatment with LUM-IVA. Visits were scheduled on the first day of treatment and every 3 months evaluating: symptoms, Body Mass Index (BMI), spirometry, laboratory tests and Quality of life. At baseline and at 12 months, the patients underwent sweat test, oral glucose tolerance test (OGTT), chest CT and dual-energy X-ray absorptiometry (DEXA).

DETAILED DESCRIPTION:
Introduction Cystic fibrosis (CF) is a genetic multisystem disease that is characterized by pancreatic insufficiency (PI) and chronic airway infections associated with loss of lung function, repeated pulmonary exacerbations (PEx), and ultimately, respiratory failure. F508del, the deletion of a single amino acid, is the most common mutation that causes CF. In July 2015, the U.S. Food and Drug Administration approved the combination Lumacaftor/Ivacaftor (Orkambi®, Vertex pharmaceuticals) for use in patients with CF homozygous for the F508del mutation. Briefly, this combination of a corrector (Lumacaftor) and potentiator (Ivacaftor) partially restores the activity of the membranous CF transmembrane regulator (CFTR) protein. Lumacaftor improves the processing of F508del CFTR and its transport to the cell surface, while Ivacaftor increases the probability for the channel to be open and its transport of chloride. In clinical trials, treatment with Lumacaftor-Ivacaftor (LUM-IVA) in individuals homozygous for F508del led to an increase in lung function, weight, and a significant reduction in the frequency of PEx and CF-related hospitalizations.

Extra-pulmonary complications are common in CF. Of these, CF-related diabetes (CFRD) is one of the worst prognostic factors. In people with gating mutations responsive to Ivacaftor, treatment was associated with an improvement in insulin secretion after glucose challenge.

Another important extra-pulmonary complication is CF bone disease (CFBD), characterized by low bone mineral density. Osteopenia and fractures are noted among 50-75% of patients diagnosed with CF. The reasons for those pathologies are malabsorption of fat soluble vitamins, a complex abnormality of sex hormone composition, primary CFTR dysfunction, chronic infection and inflammation, and low levels of bone-building exercise resulting from advanced respiratory compromise. It is well known that growth and sexual development is delayed in CF patients, due in part to nutritional deficiencies and the severity of their chronic lung disease. These delays are accompanied by low levels of sex hormones: luteinizing hormone (LH) and follicle-stimulating hormone (FSH).

The aim of the current study was to evaluate endocrine pancreatic function, bone metabolism and respiratory changes through the first year of LUM-IVA treatment in adult patients.

Materials and methods Study design and participants The study was a prospective, single center, observational real-world study on F508del homozygous adult CF patients, who commenced treatment with LUM-IVA and were followed for a year. Pregnant and nursing females; solid organ or hematological transplant recipients; alcohol or drug abusers; patients with an acute upper or lower respiratory infection, and those with PEx or changes in therapy for pulmonary disease within 28 days before Day 1 (first dose of study drug) were excluded.

All subjects received 400 mg Lumacaftor /250 mg Ivacaftor (LUM-IVA) fixed-dose combination film coated tablets for oral administration every12 hours. All participants remained on their pre-study stable CF medication regimen through the year. They were followed in the CF Center at Carmel Medical Center, Haifa, Israel between 2016 and 2019. The institutional board reviewed and approved the study protocol. All patients provided written informed consent.

Study period Screening period was from day -28 through day -1. Treatment period was from day 1 (first dose of study drug) through 12 months ± 7 days. Five clinic visits were carried out on day 1 and at weeks 12, 24, 36 and 48 (± 7 days).

At screening (V0) and at 12 months (V5) the patients underwent a sweat test, Oral glucose tolerance test (OGTT) in patients without CF related diabetes (CFRD), chest computed tomography (CT) and a bone density evaluation using Dual-energy x-ray absorptiometry (DEXA). Evaluations performed during each visit included: recording of CF-related symptoms, treatments, physical examination, vital signs, body mass index (BMI) measurements, pulmonary function tests (PFT), laboratory tests, sputum culture and disease-specific quality of life evaluation using the Cystic Fibrosis Questionnaire-Revised (CFQR).

Study assessments The primary endpoint was the absolute change from baseline through 12 months in the percentage of predicted Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and forced expiratory flow between 25-75 (FEF25-75). Spirometry was performed in accordance with the American Thoracic Society/ European Respiratory Society (ATS/ERS ) Task Force, using a KoKo® spirometer (n-Spire Healthcare, Inc., Longmont CO, USA).

Key secondary endpoints included the absolute and relative change from baseline through 12 months in (1) metabolic factors, including BMI, OGTT (75g of glucose were ingested orally, and glucose, insulin & c-peptide were examined at the time of ingestion, 1 hour and 2 hours later), Albumin and HbA1C; (2) bone health factors including parathyroid hormone (PTH), Alkaline phosphatase, , Phosphor, and Calcium levels; A, D, E vitamin levels, Urine Ca/Cr ratio; and DEXA scans (3) Hormonal factors including; luteinizing hormone (LH), follicle stimulating hormone (FSH), Testosterone and Estradiol levels; and (4) evaluation of CFTR function through concentration of sweat chloride Additional evaluations included (1) chest CT scans that were performed and scored using the Bhalla scoring method by a radiologist-investigator (the total score ranges from 9 to 25, with a higher score indicating more severe structural lung changes); (2) The patient-reported CFQ-R respiratory domain score (scores range from 0 to 100, with higher scores indicating a better quality of life and 4 points considered to be a minimal clinically important difference) (3) safety parameters (electrolytes, liver and kidney function test, coagulation function) and (3) pulmonary exacerbations (PEx). A PEx was defined as a deterioration in respiratory symptoms that led to a change in treatment. Each PEx was counted as a separate event, and the number of PEx in the year prior to commencing treatment with LUM-IVA was compared to PEx in the year on the treatment. We documented: number of exacerbations, oral vs. intravenous antibiotic treatment, hospitalizations, presence of fever >38°C, laboratory parameters (white blood cells count [WBC], absolute neutrophil count [ANC], C-reactive protein [CRP] at PEx start in hospitalized patients), sputum culture results and time to next PEx.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following inclusion criteria will be eligible for this study:

  1. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, and other study procedures.
  2. Subjects (males and females), will be aged 18 years or older
  3. Confirmed diagnosis of CF
  4. Homozygous for the F508del-CFTR mutation.
  5. Willing to remain on a stable CF medication regimen through 12 months.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible for this study:

  1. History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.

     For example:

     • History of cirrhosis with portal hypertension, and/or history of risk factors for Torsade de Pointes (e.g., familial long QT syndrome, hypokalemia, heart failure, left ventricular hypertrophy, bradycardia, myocardial infarction, cardiomyopathy, history of arrhythmia [ventricular and atrial fibrillation]), obesity, acute neurologic events.
  2. Any of the following abnormal laboratory values at Screening:

     * Abnormal liver function defined as any 2 or more of the following: ≥3 × upper limit of normal (ULN) aspartate aminotransferase (AST), ≥3 × ULN alanine aminotransferase (ALT), ≥3 × ULN gamma-glutamyl transpeptidase (GGT), ≥3 × ULN alkaline phosphatase (ALP), or ≥2 × ULN total bilirubin
     * Abnormal liver function defined as any increase of ≥5 × ULN AST or ALT
     * Abnormal renal function defined as glomerular filtration rate ≤50 mL/min/1.73 m2
  3. An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1 (first dose of study drug).
  4. History of solid organ or hematological transplantation.
  5. History or evidence of cataract, lens opacity, Y-suture, or lamellar rings determined to be clinically significant by the ophthalmologist during the ophthalmologic examination during the Screening Period.
  6. History of alcohol or drug abuse in the past year, including but not limited to cannabis, cocaine, and opiates, as deemed by the investigator.
  7. Pregnant or nursing females: Females of childbearing potential must have a negative pregnancy test at Screening and Day 1.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: F508del homozygous adult CF patients, who commenced treatment with LUM-IVA in a single center
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Pulmonary function tests | 1 year
  the absolute change from baseline through 12 months in the percentage of predicted Forced expiratory volume in 1 second (FEV1).

SECONDARY OUTCOMES:
BMI | 1 year
  weight and height will be combined to report BMI in kg/m^2
bone parameters | 1 year
  Alkaline phosphatase - absolute and relative change from baseline ( every 3 months under treatment)
bone health factors | 1 year
  DEXA scans
Additional Pulmonary function tests | 1 year
  the absolute change from baseline through 12 months in the percentage of predicted forced expiratory flow between 25-75 (FEF25-75).
Glucose metabolism | The change between 12 months (under treatment) to screening
  OGTT (75g of glucose were ingested orally, and glucose was examined at the time of ingestion, 1 hour and 2 hours later)- we will report the glucose parameter of OGTT test.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Yaacoby-Bianu, MD, Principal Investigator — Carmel Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758